CLINICAL TRIAL: NCT03338712
Title: Micro-RNA Expression Profiles in Localised Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigators no longer in business
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: mi-RNA-PCa
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recurrence free survival The patients will be followed in regular time intervals in accordance with the EAU-Guidelines (2010) and the S-3 Guideline for Prostate cancer of the German Urological Association. Data will be updated once yearly for until death.

ELIGIBILITY:
Inclusion Criteria:

* 35 Years to 80 Years
* Male
* Patients with clinically localised high risk prostate cancer

Exclusion Criteria:

-

Ages: 35 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: * Male
  * Patients with clinically localised high risk prostate cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | Up to 120 months. From date of inclusion until date of death from any cause
  The patients will be followed in regular time intervals in accordance with the EAU-Guidelines (2010) and the S-3 Guideline for Prostate cancer of the German Urological Association.

SECONDARY OUTCOMES:
Cancer specific survival | Up to 120 months. From date of inclusion until date of death from any cause
  Cancer specific survival

IPD SHARING:
Plan to Share IPD: No